CLINICAL TRIAL: NCT00114153
Title: Phase I Trial of Induction Paraplatin® and Xeloda® Followed by Concurrent Paraplatin and Xeloda With Intensity Modulated Radiotherapy for Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Carboplatin, Capecitabine, and Radiation Therapy in Treating Patients With Stage III or Stage IV Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000432949; UVACC-HIC-10519; UVACC-27402; BMS-UVACC-HIC-10519
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2007-04

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Capecitabine; Carboplatin; Radiotherapy

INTERVENTIONS:
Drug: capecitabine
Drug: carboplatin
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of capecitabine when given together with carboplatin followed by radiation therapy in treating patients with stage III or stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) of capecitabine when administered with carboplatin as induction chemotherapy in patients with stage III-IVB squamous cell carcinoma of the head and neck.
* Determine the MTD of capecitabine when administered with concurrent carboplatin and intensity-modulated radiotherapy in these patients.
* Determine the toxicity of this regimen in these patients.

Secondary

* Determine, preliminarily, tumor response in patients treated with this regimen.
* Determine the quality of life of patients treated with this regimen.

OUTLINE: This is a dose-escalation study of capecitabine.

* Induction chemotherapy: Patients receive carboplatin IV on days 1, 8, 15, 22, 29, and 36 and oral capecitabine twice daily on days 1-14 and 22-35.
* Concurrent chemoradiotherapy: Beginning 2 weeks after completion of induction chemotherapy, patients receive carboplatin and capecitabine as in induction chemotherapy. Patients also undergo intensity-modulated radiotherapy (IMRT) once daily on days 1-5, 8-12, 15-19, 22-26, and 29-33 and non-IMRT boost once daily on days 36-40 and 43-47.

Treatment continues in the absence of disease progression or unacceptable toxicity.

Within 4-8 weeks after completion of concurrent chemoradiotherapy, patients who achieve a clinical complete response or who are medically operable with resectable persistent or recurrent disease undergo neck dissection (salvage surgery).

Cohorts of 3-6 patients receive escalating doses of capecitabine (during both induction chemotherapy and concurrent chemoradiotherapy) until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Quality of life is assessed at baseline, after completion of induction chemotherapy, and then at 1 week and 3, 6, and 12 months after completion of concurrent chemoradiotherapy.

After completion of study therapy, patients are followed monthly for 3 months and then every 3 months for 1 year.

PROJECTED ACCRUAL: Approximately 6-48 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck, including 1 of the following types:

  * Oral cavity
  * Oropharynx
  * Hypopharynx
* Clinical stage III-IVB (T2-T4, N0-N3, M0) disease
* Measurable disease by physical exam, endoscopy, and/or CT scan or MRI

  * Residual measurable disease after fine needle aspiration, core needle biopsy, or incisional or excisional biopsy of the primary tumor
* No evidence of distant metastases (M1)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 9 g/dL
* No uncontrolled coagulopathy

Hepatic

* AST < 2 times normal
* Alkaline phosphatase < 2 times normal
* Bilirubin normal

Renal

* Creatinine < 2.0 mg/dL OR
* Creatinine clearance > 50 mL/min

Cardiovascular

* No congestive heart failure
* No symptomatic coronary artery disease
* No uncontrolled cardiac arrhythmias
* No myocardial infarction within the past year
* No other clinically significant cardiac disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 30 days after completion of study treatment
* Nutritional and general physical condition must be compatible with proposed study treatment
* Mentally reliable
* No pre-existing peripheral neuropathy > grade 1
* No history of hypersensitivity to fluorouracil, capecitabine, or carboplatin
* No active infection
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* No major medical, psychiatric, or neurologic illness that would preclude study participation or giving informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 5 years since prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for head and neck tumor
* No prior radiotherapy to the region of planned study radiotherapy fields

Surgery

* Recovered from prior surgery

  * No unhealed surgical wounds

Other

* More than 4 weeks since prior investigational drugs
* No concurrent warfarin, diphenylhydantoin, or fluconazole unless willing to undergo careful monitoring and appropriate dose adjustments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2003-06

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Y. Thomas, MD, Principal Investigator — University of Virginia; Paul W. Read, MD, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Cancer Center at UV Health System, Charlottesville, Virginia, United States

REFERENCES:
- [Result] Thomas CY, Read P, Petroni G, Reibel J, Levine PA. Phase I study of capecitabine, carboplatin and intensity-modulated radiation therapy for head and neck cancer. Anticancer Res. 2009 Jul;29(7):2869-73. PMID 19596976